CLINICAL TRIAL: NCT04584944
Title: Appendicular Skeletal Muscle Mass Adult Reference Measurements in Greek Population
Brief Title: Appendicular Skeletal Muscle Mass Study
Acronym: SmmS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henry Dunant Hospital Center (Other)
Responsible Party: Sponsor
Other Study IDs: 3080234A
Record Dates: First submitted 2020-09-03; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Public Health; Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Absorptiometry, Photon; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy adult men: Healthy young men, 20- 44 years old
  Interventions: Radiation: Dual energy X-ray absorptiometry
- Healthy adult women: Healthy young women, 20- 44 years old
  Interventions: Radiation: Dual energy X-ray absorptiometry

INTERVENTIONS:
Radiation: Dual energy X-ray absorptiometry — Evaluation of the appendicular muscle mass of the limbs will be performed by Dual-Energy X-ray Absorptiometry, using a QDR 4500. Body composition analysis will also be evaluated with TANITA Body Composition Analyzer device,model BC-418MA. Bioelectrical Impedance Analysis measures the body composition using a constant power source (high frequency current 50kHz, 90 μA).
  Muscle mass is also going to be measured by using ultrasound -U/S. It measures basic parameters such as muscle volume and spectrum length through the B-Mode imaging with Linear 7-12MHz frequency heads that can reliably determine the thickness and transverse incisions of the superficial muscular Groups.
  Other Names: Bioelectrical Impedance Analysis; Ultrasound

SUMMARY:
There is a lot of discussion concerning the normal cut-off points of skeletal mass among different populations worldwide. Genetic and environmental differences most probably lead to different measurements. Defining muscle mass in healthy young adults in Greece will provide information that can be used to determine normal ranges of muscle mass of both sexes and consequently define sarcopenia.

The aim of the study is to define appendicular skeletal muscle mass reference measurements in healthy young adults in Greece. These values can be used to determine sarcopenia cut-offs according to recommendations.

DETAILED DESCRIPTION:
Introduction

The reduction of muscle mass in humans is obvious after the age of fifty, with a reduction rate of 3-8% every ten years. The rate of loss accelerates with chronic diseases, sedentary lifestyle, low physical activity, nutritional, environmental and socioeconomic factors .

Sarcopenia has been officially recognized as a disease according to World Health Organization. European Working Group on Sarcopenia in Older People 2 has revised the definition and diagnostic criteria of sarcopenia aiming to encourage more research in the field. In Greece, there are no reference values for muscle strength and muscle mass. Defining these values will permit the investigators to provide a tool that will help to establish country - specific measurements of sarcopenia in Greek population.

Study population-Methods

The study site will be the Outpatient Geriatric Assessment Unit and the Radiology Department of Henry Dunant Hospital Centre, in Athens-Greece.

The study population will be healthy adults that meet the inclusion criteria. The recruitment will be performed using the snowball sampling technique (for instance, through printed material, the marketing department of the hospital, social media, advertising banners, etc.). Stratified random sampling technique will be used to achieve a representative sample size.

Evaluation of the appendicular muscle mass of the limbs will be performed by Dual-Energy X-ray Absorptiometry, using a QDR-4500 A fan Beam densitometer (Hologic, Inc., Bedford, MA). Hologic Discovery W configured with software version 12.1 (Hologic, Bedford, MA).

Body composition analysis will be evaluated with TANITA Body Composition Analyzer device,model BC-418MA. Analysis concerns calculation of body consistency (body fat mass, lean mass water and predicted muscle mass) using Bioelectric Impedance Analysis. Bioelectric Impedance Analysis measures the body composition using a constant power source (high frequency current 50kHz, 90 μA).

Muscle mass will also be measured by ultrasound -U/S. U/S determines the thickness and transverse incisions of a superficial muscle group. It can measure basic parameters such as muscle volume and spectrum length through the B-Mode imaging with Linear 7-12MHz frequency heads that can reliably determine the thickness and transverse incisions of the superficial muscular Groups.

Statistical analysis

It will be performed using the Statistical Package for the Social Sciences -SPSS Version 26.0 (IBM), and R Version 3.6.2.

Descriptive statistics will be presented in percentage proportions, mean values and Standard Deviations (SD) of the variables. In addition, Z-score will be calculated (e.g. Dual-energy X-ray absorptiometry , Bone Mineral density, Dual-energy X-ray absorptiometry % fat, etc.) and T-score ± 2 standard deviations.

Chi-square - χ2 tests or non-parametric tests will be produced to compare qualitative variables. T-test, Analysis of Variance- ANOVA and non-parametric tests will be used in the statistical analysis of quantitative variables within the categories of qualitative variables.

Approval

The protocol has been approved by the Scientific Committee of the Henry Dunant Hospital Centre, in Athens -Greece, and is in accordance with the Code of Ethics of the World Organization for Medical Sciences (CIOMS) as formulated in the Helsinki Declaration on Biological Research.

Informed consent

All participants will be informed in written for the purpose of the research, and the way their personal data are processed (name, address, telephone, e-mail), under the provisions of 2016/679 according to the General Data Protection Regulation (GDPR).

The consent form will describe the legal and transparent way of processing their data, stating the specific purpose for data collection, as well as information about storage of their data. It will also contain a written description of the rights of the participants concerning their data and their ability to revoke consent for the processing of their data. The processing, transfer and storage of data, will also be described, as well as who will have access to their data, and how long the data will be stored for.

Finally, all participants will sign the written informed consent and confidentiality form.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Greek young adults (20 - 44 years old), with Caucasian characteristics.
2. Able to read and write in Greek language.

Exclusion Criteria:

1. Chronic diseases, such as, heart diseases, type II diabetes mellitus and autoimmune diseases.
2. Hyperthyroidism or hypothyroidism (persons with normal thyroid function for six months are included).
3. Malignancies.
4. Seizures of epilepsy, neurodegenerative diseases.
5. Asthma and/or chronic respiratory pulmonary disease-Chronic Obstructive Pulmonary Disease.
6. Metal prefixes.
7. Pacemaker.
8. Systematic medication intake (such as hypolipemic drugs, antihypertensive drugs, antidepressants, glucocorticoids and any other hormonal treatment).
9. Protein formulations and anabolic intake.
10. Hormone intake (testosterone, estrogen, contraceptive, growth hormone, dehydroepiandrosterone.
11. Professional athletes and people with intense physical activity, intensive exercise with weights, long-distance runners (Marathons).
12. Substance use or abuse (cocaine, heroin, amphetamines).
13. Pregnancy.
14. History of hospitalization in Intensive Care Unit
15. History of serious injury
16. Considerable body weight alterations during the previous year (increase or decrease)
17. History of Bariatric surgery
18. Any dietary restriction due to disease (sprue), choice (vegan), or eating disorder (anorexia nervosa).

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gender identity
Study Population: The study population will be healthy adults that meet the inclusion criteria and can have access to the study site. The recruitment will be performed using the snowball sampling technique (for instance, through printed material, the marketing department of the hospital, social media (Facebook/Instagram/Twitter), advertising banners, etc.). We will also invite participants from nearby academic institutions, organizations, municipalities, etc. It is foreseen to include 500 participants in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Appendicular skeletal muscle mass reference measurements of healthy young adults in Greece | 01/06/2022
  Measurements of appendicular skeletal muscle mass of healthy young adults in Greece that will be used to define sarcopenia in older adults and as normative values.
Define reference measurements for muscle strength. | 01/06/2022
  Reference measurements for hand grip
Define reference measurements for muscle performance | 01/06/2022
  Reference measurements for walking speed

SECONDARY OUTCOMES:
Correlations between the different tools used to measure muscle mass | 01/06/2022
  Investigate accuracy and potential differences between the different techniques used to measure muscle mass.
Correlation of muscle mass with demographic characteristics | 01/06/2022
  Investigate correlation of muscle mass with demographic characteristics of the studied population
Correlation of bone mass with demographic characteristics | 01/06/2022
  Investigate correlation of bone mass with demographic characteristics of the studied population.
Correlation of fat mass with demographic characteristics | 01/06/2022
  Investigate correlation of fat mass with demographic characteristics of the studied population.
Correlation of adherence to Mediterranean diet with muscle mass | 01/06/2022
  Investigate potential correlation of adherence to Mediterranean diet with muscle mass.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia Koutsouri, Study Chair — Head of the Outpatient Geriatric Assessment Unit
Locations (1):
- Henry Dunant Hospital Center, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Result] Buckinx F, Landi F, Cesari M, Fielding RA, Visser M, Engelke K, Maggi S, Dennison E, Al-Daghri NM, Allepaerts S, Bauer J, Bautmans I, Brandi ML, Bruyere O, Cederholm T, Cerreta F, Cherubini A, Cooper C, Cruz-Jentoft A, McCloskey E, Dawson-Hughes B, Kaufman JM, Laslop A, Petermans J, Reginster JY, Rizzoli R, Robinson S, Rolland Y, Rueda R, Vellas B, Kanis JA. Pitfalls in the measurement of muscle mass: a need for a reference standard. J Cachexia Sarcopenia Muscle. 2018 Apr;9(2):269-278. doi: 10.1002/jcsm.12268. Epub 2018 Jan 19. PMID 29349935
- [Result] Wong AK. A Comparison of Peripheral Imaging Technologies for Bone and Muscle Quantification: a Mixed Methods Clinical Review. Curr Osteoporos Rep. 2016 Dec;14(6):359-373. doi: 10.1007/s11914-016-0334-z. PMID 27796924
- [Result] Mijnarends DM, Luiking YC, Halfens RJG, Evers SMAA, Lenaerts ELA, Verlaan S, Wallace M, Schols JMGA, Meijers JMM. Muscle, Health and Costs: A Glance at their Relationship. J Nutr Health Aging. 2018;22(7):766-773. doi: 10.1007/s12603-018-1058-9. PMID 30080217
- [Result] Schaap LA, van Schoor NM, Lips P, Visser M. Associations of Sarcopenia Definitions, and Their Components, With the Incidence of Recurrent Falling and Fractures: The Longitudinal Aging Study Amsterdam. J Gerontol A Biol Sci Med Sci. 2018 Aug 10;73(9):1199-1204. doi: 10.1093/gerona/glx245. PMID 29300839
- [Result] Malmstrom TK, Miller DK, Simonsick EM, Ferrucci L, Morley JE. SARC-F: a symptom score to predict persons with sarcopenia at risk for poor functional outcomes. J Cachexia Sarcopenia Muscle. 2016 Mar;7(1):28-36. doi: 10.1002/jcsm.12048. Epub 2015 Jul 7. PMID 27066316
- [Result] Chang KV, Hsu TH, Wu WT, Huang KC, Han DS. Association Between Sarcopenia and Cognitive Impairment: A Systematic Review and Meta-Analysis. J Am Med Dir Assoc. 2016 Dec 1;17(12):1164.e7-1164.e15. doi: 10.1016/j.jamda.2016.09.013. Epub 2016 Nov 2. PMID 27816484
- [Result] Antunes AC, Araujo DA, Verissimo MT, Amaral TF. Sarcopenia and hospitalisation costs in older adults: a cross-sectional study. Nutr Diet. 2017 Feb;74(1):46-50. doi: 10.1111/1747-0080.12287. Epub 2016 Jun 13. PMID 28731551
- [Result] Beaudart C, Rizzoli R, Bruyere O, Reginster JY, Biver E. Sarcopenia: burden and challenges for public health. Arch Public Health. 2014 Dec 18;72(1):45. doi: 10.1186/2049-3258-72-45. eCollection 2014. PMID 25810912
- [Result] Lourenco RA, Perez-Zepeda M, Gutierrez-Robledo L, Garcia-Garcia FJ, Rodriguez Manas L. Performance of the European Working Group on Sarcopenia in Older People algorithm in screening older adults for muscle mass assessment. Age Ageing. 2015 Mar;44(2):334-8. doi: 10.1093/ageing/afu192. Epub 2014 Dec 23. PMID 25539836
- [Result] Panagiotakos DB, Pitsavos C, Stefanadis C. Dietary patterns: a Mediterranean diet score and its relation to clinical and biological markers of cardiovascular disease risk. Nutr Metab Cardiovasc Dis. 2006 Dec;16(8):559-68. doi: 10.1016/j.numecd.2005.08.006. Epub 2006 Feb 9. PMID 17126772
- [Derived] Soulis G, Zigkiri E, Perkisas S, Antoniou K, Maniati A, Galanos A, Georgiadis E, Koutsouri A. Muscle Mass Reference Values of Greek Adult Population: A Cross-Sectional Study for Sarcopenia Definition in Greece. J Musculoskelet Neuronal Interact. 2025 Dec 1;25(4):422-429. doi: 10.22540/JMNI-25-422. PMID 41324213